CLINICAL TRIAL: NCT05665686
Title: Investigation of the Efficacy of Different Treatment Approaches on Sexual Health in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, physiotherapist PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sexual Health
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Floor Disorders
Keywords: woman's health; exercise
MeSH Terms: conditions — Pelvic Floor Disorders; Motor Activity | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Group (Experimental): Sexual Information and Advice to Individuals Individuals in both groups will be given training on sexuality. Male and female sexual situation, orgasm, male and female anatomical structures will be explained. At the same time, information will be given about the pelvic floor muscles, their function and their importance in sexual life.
  Interventions: Device: Relaxation training with device
- home exercise (Active Comparator): A home exercise program including pelvic floor relaxation exercises in different positions will be created for individuals in both groups and self-myofascial massages will be taught. At the same time, information will be given about the pelvic floor muscles, their function and their importance in sexual life.
  Interventions: Other: Home Exercise

INTERVENTIONS:
Device: Relaxation training with device — Relaxation training will be applied with the device.
  Arms: Device Group
Other: Home Exercise — An exercise application including home exercise programs will be performed for six weeks.
  Arms: home exercise

SUMMARY:
Sexual health is one of the important factors affecting the quality of life and general health of individuals.

Sexual life, with its personal and social aspects, is an inseparable part of the human being in general. It is one of the most important factors in human life and happiness, especially in family life.

Sexuality positively integrates and enriches the somatic, emotional, intellectual and social aspects of individuals, and develops a personality, communication and love.

The concepts of sexuality and sexual health have long been considered taboo. This situation negatively affects rehabilitation strategies. Studies are known to have sexual problems in women more than men.

DETAILED DESCRIPTION:
There are many factors that affect sexual function. In the etiology of female sexual dysfunction; neurogenic, vascular, hormonal, musculogenic and psychogenic factors are included. If female sexual dysfunction causes distress, it negatively affects women's quality of life. The repetition of problems related to sexual response, pain, orgasm and desire, which cause interpersonal problems and discomfort, creates a complex problem.

Pelvic floor muscles are known to play an important role in sexual function as they are responsible for involuntary rhythmic contractions during orgasm and vaginal sensation during intercourse. Studies have reported that pelvic floor disorders affect one-third of adult women and significantly reduce their quality of life. Different treatment methods applied to the pelvic floor muscles increase the level of muscle strength and muscle activation. Increasing pelvic floor muscle strength affects individuals' sexual life positively and reduces the problems encountered. Conservative treatment modalities include exercises for the pelvic floor muscles, functional electrical stimulation, and surface electromyography. Exercise practices are one of the important approaches that strengthen the pelvic floor muscles.

These exercise approaches can be given in the form of home exercise applications, as well as device-assisted applications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 and over
* Having an active sex life

Exclusion Criteria:

* Latex allergy
* Other allergies in the pelvic area
* Vaginal or urinary tract infection
* Gynecological cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Scale | six weeks
  This scale was developed by Rosen et al. It has been developed by in the United States of America and its main purpose is to address female sexual function in a multifaceted manner. It has been shown to be a valid and reliable diagnostic tool in analyzing sexual functions in Turkish women. FSFI; It consists of 19 questions in total. Scale; There are 6 sub-dimensions: desire, arousal, lubrication, orgasm, satisfaction and pain. Each item is scored from zero to 5. Accordingly, the highest raw score that can be obtained from the scale is 95.0 and the lowest raw score is 4.0.
Female Sexual Stress Scale | six weeks
  This scale was first developed in 2002 in the United States by Derogatis, Pyke, McCormack, Hunter, and Harding to assess women with sexual dysfunction. When filling out the scale, women are asked to describe the frequency of discomfort with the sexual problem they have experienced in the last 30 days. In the society where this 13-item 5-point Likert-type scale was developed, women who score 11 and above are considered to have sexual disorders.
Surface electromyography | six weeks
  With the help of this measurement technique, which contains important information about the contraction of our body muscles, it is checked which muscles are activated in which movement.
  In our study, muscle activation evaluation will be made with the evaluation of the pelvic floor muscles.

SECONDARY OUTCOMES:
Sexual Life Quality Scale- Female: | six weeks
  Each item is expected to be answered by considering the sexual life in the last four weeks. Each question is scored between 1 and 6 in the scoring of the scale. The range of points that can be obtained from the scale is between 18 and 108. A high score from the scale indicates that the quality of sexual life is good.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Salazar de Pablo G, De Micheli A, Nieman DH, Correll CU, Kessing LV, Pfennig A, Bechdolf A, Borgwardt S, Arango C, van Amelsvoort T, Vieta E, Solmi M, Oliver D, Catalan A, Verdino V, Di Maggio L, Bonoldi I, Vaquerizo-Serrano J, Baccaredda Boy O, Provenzani U, Ruzzi F, Calorio F, Nosari G, Di Marco B, Famularo I, Molteni S, Filosi E, Mensi M, Balottin U, Politi P, Shin JI, Fusar-Poli P. Universal and selective interventions to promote good mental health in young people: Systematic review and meta-analysis. Eur Neuropsychopharmacol. 2020 Dec;41:28-39. doi: 10.1016/j.euroneuro.2020.10.007. Epub 2020 Nov 6. PMID 33162291